CLINICAL TRIAL: NCT03268928
Title: Evaluating the Impact of Story Starters on Children's Language Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Julian Pine (Other)
Responsible Party: Sponsor-Investigator, Julian Pine, Professor, University of Liverpool
Organization: University of Liverpool (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1869
Record Dates: First submitted 2017-08-25; First posted 2017-08-31 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2018-05

CONDITIONS: Language Development
Keywords: Shared Book Reading; Language Development; Syntax; Vocabulary; Phonological Awareness; Young Children; Randomised Control Trial; Language Intervention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Story Starters Intervention (Experimental): Children will receive the the Story Starters intervention for six months. Each child will be visited by a trained Story Starter volunteer twice a week while the child is in preschool. The sessions will last 20 minutes and in each session the Story Starter volunteer and child will read books and play with toys. The Story Starter volunteers will keep a record of the number of sessions each child attends.
  Each child will receive one new book per month delivered to their home address by Dolly Parton's Imagination Library.
  Interventions: Behavioral: Story Starters Intervention
- Wait-list Control (Other): Children in the wait-list control arm will continue to attend preschool as normal during the randomised controlled trial (RCT) and will receive the Story Starters intervention after the RCT has finished.
  Each child will receive one new book per month delivered to their home address by Dolly Parton's Imagination Library.
  Interventions: Behavioral: Wait-list Control

INTERVENTIONS:
Behavioral: Story Starters Intervention — Shared reading intervention
  Arms: Story Starters Intervention
Behavioral: Wait-list Control — Wait-list control
  Arms: Wait-list Control

SUMMARY:
The aim of this project is to evaluate whether Beanstalk's 'Story Starters' intervention is effective in boosting vocabulary and grammatical development in young children.

DETAILED DESCRIPTION:
Children who read regularly with their parents or carers tend to learn language faster, enter school with a larger vocabulary of words and become more successful readers in school. Because of this, local authorities often commission services to promote family-based shared book reading. However, recent studies suggest that shared reading interventions work less effectively for children from disadvantaged backgrounds than originally thought, particularly when their parents have lower levels of education. This means that there is a danger that the benefits of shared reading will be restricted to children from more affluent homes and not get through to those who need them most. To solve this problem, there is a need to develop a better understanding of how reading interventions work and to evaluate existing shared reading interventions to determine whether they are effective in promoting young children's language development.

The aim of this project is to evaluate whether Beanstalk's 'Story Starters' intervention is effective in boosting vocabulary and grammatical development in young children. Story Starters is a reading intervention delivered by Beanstalk, a national children's literacy charity committed to ensuring no child faces the severe consequences of illiteracy. Beanstalk trains volunteers to provide caring and fun one-to-one support to disadvantaged children aged 3 and 4 in local nurseries, aiding their language development.

The project will compare the effects of the 'Story Starters' intervention against a wait-list control group. Children in the intervention group will receive the Story Starters intervention, delivered by a trained Beanstalk volunteer, at their preschool for six months. The trained volunteer will visit the child twice a week and deliver a one-to-one 20 minute book reading and play session. Children in the intervention group will also receive a new book each month which will be sent to their home address by Dolly Parton's Imagination Library.

Children in the wait list control group will also receive a new book each month from Dolly Parton's Imagination Library but they will not receive the 'Story Starters' intervention until after the project has ended.

ELIGIBILITY:
Inclusion Criteria:

All families will be included unless they fit the exclusion criteria

Exclusion Criteria:

* Children born before 37 weeks gestation (premature)
* Children who weighed less than 5lb 9oz at birth (low birth weight)
* Children who have had an ear infection/glue ear for longer than 3 months, 4-6 ear infections within a 6 month period or another identified hearing problem (e.g. at newborn hearing screening)
* Children with an identified developmental disability (e.g. Cerebral Palsy, Autism Spectrum Disorder, Fragile X syndrome, Muscular dystrophy, Di George syndrome, Down's syndrome, Williams syndrome)
* Children with a hearing or visual impairment
* Children who hear another language (not English) for 1 day or more in a typical week (please note that this also excludes children of parents who do not speak English)
* Children whose parents have a learning disability which puts their children at risk of language delay and excludes the parents from giving informed consent on their own and on their children's behalf.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 198 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Change in baseline language skills - CELF | Baseline, 6 months and 12 months
  The Clinical Evaluation of Language Fundamentals - Preschool 2 United Kingdom (CELF Preschool-2) will be administered. This is a published standardized measure of the language knowledge of individual children. The investigators will use three subtests to calculate each child's core language score. The three subtests measure knowledge of sentence structure, knowledge of word structure and expressive vocabulary.
Change in baseline receptive vocabulary | Baseline, 6 months and 12 months
  The British Picture Vocabulary Scale (BPVS) will be administered. This is a published standardised measure and will be used to measure receptive vocabulary of individual children.
Change in baseline phonological awareness | Baseline, 6 months and 12 months
  The full Preschool Inventory of Phonological Awareness (PIPA) will be administered. This is a published standardised measure of phonological awareness of individual children. The investigators will use the PIPA to measure, rhyme awareness, syllable segmentation, alliteration awareness, phoneme isolation, phoneme segmentation and letter knowledge.
Change in baseline language skills - the WellComm Screening tool | Baseline, 6 months and 12 months
  The WellComm Screening Tool will be administered. This is a published measure of language skills of individual children. The investigators will use the WellComm to measure expressive and receptive language skills.

SECONDARY OUTCOMES:
Fidelity to the intervention by the Beanstalk volunteer | 6 months
  Video recordings of the trained Beanstalk volunteers delivering 'Story Starter' sessions will be analysed to measure fidelity to the intervention and presence of target book reading behaviours. This will include coding for the presence of Dialogic book reading behaviours (prompting, evaluating, expanding and repeating). This will allow measurement of whether the volunteer adheres to the Story Starter intervention.
Child engagement | 6 months
  Video recordings of the trained Beanstalk volunteers delivering 'Story Starter' sessions will be analysed to measure level of child engagement (Kucirkova, Messer & Whitelock, 2012). This will include coding rate of pointing, rate of smiles and laughs, rate of less engaged behaviours and rate of vocal activity.
Volunteer engagement | 6 months
  Video recordings of the trained Beanstalk volunteers delivering 'Story Starter' sessions will be analysed to measure level of volunteer engagement (Kucirkova, Messer & Whitelock, 2012). This will include coding rate of pointing, rate of smiles and laughs, rate of less engaged behaviours and rate of vocal activity.

CONTACTS AND LOCATIONS:
Overall Officials: Julian Pine, PhD, Principal Investigator — The University of Liverpool
Locations (1):
- Liverpool Language Lab at the University of Liverpool, Liverpool, Merseyside, United Kingdom

REFERENCES:
- [Background] Kucirkova, N, Messer, D, Whitelock, D. Parents reading with their toddlers: the role of personalisation in book engagement. Journal of Early Childhood Literacy, 13(4): 445-470, 2012
- [Background] Bus AG, van IJzendoorn MH, Pellegrini AD. Joint book reading makes for success in learning to read: A meta-analysis on intergenerational transmission of literacy. Review of Educational Research, 65: 1-21, 1995.
- [Background] Mol SE, Bus AG, de Jong MT, Smeets DJH. Added value of dialogic parent-child book readings: A meta-analysis. Early Education and Development, 19: 7-26, 2008